CLINICAL TRIAL: NCT04352179
Title: Evaluation of Patient Education Simulations to Promote Health and Wellness in Patients With Chronic Disease
Brief Title: Evaluation of Patient Education Simulations to Promote Health and Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-00460
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Chronic Disease
Keywords: Lifestyle
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Education Simulation (Experimental): All participants will have access to the virtual education simulations.
  Interventions: Behavioral: Virtual Education Simulation

INTERVENTIONS:
Behavioral: Virtual Education Simulation — The simulations will be developed using Kognito's proprietary Conversation Platform.
  In this pilot study, the simulations will be a bundle of four topic-based conversations with Linda, a virtual peer with a chronic disease. The four wellness topics are:
  1. Fitness & Nutrition
  2. Smoking Cessation
  3. Alcohol Use
  4. Distress & Anxiety

SUMMARY:
This pilot study will use a pre-post design to explore the utility of using virtual simulations to provide participant education and counseling for adopting healthy lifestyle behaviors (i.e., physical activity, nutrition, smoking, alcohol use, and anxiety/distress screening) to 60 participants with chronic diseases where lifestyle management is paramount to well-being and disease control (e.g., cardiovascular disease, stroke, diabetes, cancer, chronic obstructive pulmonary disease, osteoarthritis). Participants will have access to the simulations through a unique password-protected link over the course of one month. Participants will complete two study visits that are 30-60 minutes in duration each. There is also one optional telephone interview with a mental health professional. The telephone interview it estimated to be 10 minutes in duration and will be audiotapes, with participants' permission. The study surveys will be administrated at baseline, immediately following the simulation use and at one-month baseline measures. The measures will assess lifestyle behaviors related to healthy eating, physical activity, emotional health, smoking behaviors and alcohol use. Measures will also assess the psycho-social constructs of intrinsic motivation and self-efficacy. Finally, the usability of and satisfaction with the simulations will be explored through feedback surveys. The investigator will also seek permission to collect data from the patient's medical chart. Feedback will also be collected from four healthcare providers.

DETAILED DESCRIPTION:
The overarching goal of the pilot study is to assess the acceptability and potential efficacy of the participant education simulation on changes in participants with chronic diseases' lifestyle behaviors as well as motivation and self-efficacy to change.

The primary objective is to examine the acceptability (satisfaction, usability) of using virtual simulations to deliver participant education and counseling for adopting healthy lifestyle behaviors among a sample of four healthcare providers and 60 participants with chronic disease. The secondary objectives include examining changes in lifestyle behaviors (e.g., healthy eating, physical activity) one-month following the use of the participant education simulations in a sample of 60 participants with chronic disease (e.g. cancer, cardiovascular disease, diabetes, stroke, arthritis) and to explore the potential mediators (e.g. motivation and self-efficacy) of the simulation effects on the changes in participants' lifestyle behaviors.

Participants will communicate with a virtual human, Linda, by selecting from a dynamic menu of dialogue options. Once the learner chooses a dialogue option, they see the virtual human respond by providing personalized feedback and give users an opportunity to revise their choice. In this study, the simulations will be a bundle of four topic-based conversations with Linda, which include fitness and nutrition, smoking cessation, alcohol use, distress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Have a diagnosis of a chronic disease (e.g., osteoarthritis, coronary artery disease, chronic obstructive pulmonary disease, asthma, diabetes, hypertension, stroke, and congestive heart failure) as indicated by self-report or review of the electronic medical record; and
3. Receiving care within the NYU Langone Health Network (e.g., Faculty Group Practices and ambulatory care centers, NYU Winthrop Surgical Associates)

Exclusion Criteria:

1. Are unable to give informed consent
2. Refuse to participate
3. Any active terminal illness, mental incompetence, or uncontrolled psychiatric illness. These exclusions were based on the premise that the presence of any of these conditions would dominate the subject's perception of lifestyle management of their chronic disease.
4. Unable to speak and read in English. Patients that are unable to speak and read in English will be excluded from the proposed project because the simulations are being developed in English only. Once we demonstrate the initial efficacy of this tool, future simulations will be developed in languages other than English. Despite the language restrictions, no exclusion will be made based on patient racial/ethnic origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who were unsatisfied and satisfied by use of virtual simulations for education delivery and counseling | Immediately post-simulation (Day 0)
  A Usability Questionnaire will be used for participants to rate how much they agree or disagree with 14 questions as they relate to the participants' conversation with the virtual coach. Choices for each question range include: strongly disagree, somewhat disagree, somewhat agree, and strongly agree. No numerical scale is used.

SECONDARY OUTCOMES:
Change in score of Alcohol Abstinence Self-Efficacy (AASE) Scale | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  The AASE Scale consists of 40 situations that lead some people to drink. Participants mark answers which reflect how tempted they may be to drink in each situation at the present time. The answers choices range from 0 (not at all) to 4 (extremely). The range of score is 0-160. The higher the score, the higher the temptation to drink.
Score of Short Portable Mental Status Questionnaire (SPMSQ) | Baseline (Day 0)
  10 questions will be asked to the participants. All responses must be given without reference to calendar, newspaper, birth certificate, or other aid to memory. The total number of errors based on the answers to the 10 questions will be recorded as the score. The lower the score, the better. 0-2 errors = Intact Intellectual Functioning, 3-4 errors = Mild Intellectual Impairment, 5-7 errors = Moderate Intellectual Impairment, 8-10 errors = Severe Intellectual Impairment.
Change in score of Smoking Abstinence Self-Efficacy Questionnaire (SASEQ) | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  The SASEQ consists of 6 situations that lead some people to smoke. Participants mark answers which reflect how confident they feel that they will not smoke in each situation. The answer choices range from 0 (certainly) to 4 (certainly not). The range of score is 0-24.
Score of Patient Health Questionnaire-8 (PHQ-8) | Baseline (Day 0)
  PHQ-8 consists of 8 problem situations. The questionnaire asks the participants how often they have been bothered by each problem over the last 2 weeks. The total score ranges from 0-12, with categories of psychological distress being: none (0-2), mild (3-5), moderate (6-8), and severe (9-12). Therefore, the lower the score, the better.
Change in amount of days of physical activity | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  Three types of physical activity will be reported on: vigorous, moderate, and walking. Participants will report how many days they did vigorous physical activities (like heavy lifting, digging, aerobics, or fast bicycling), how many days they did moderate (carrying light loads, bicycling at a regular pace, doubles tennis), and how many days they walked for at least 10 minutes during the last 7 days.
Change in Score of Self Efficacy Fruits and Vegetables Questionnaire | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  This questionnaire consists of 10 statements. The participant must rate how confident they are about each of the statements. The responses range from 0 (not at all sure) to 3 (very sure). The total score ranges from 0-30. The higher the score, the more confident the participant is about incorporating fruits and vegetables into their lifestyle.
Change in Score of Self Efficacy Exercising Questionnaire | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  This questionnaire consists of 11 statements. The participant must rate how confident they are about each of the statements. The responses range from 0 (not at all sure) to 3 (very sure). The total score ranges from 0-30. The higher the score, the more confident the participant is about incorporating exercise into their lifestyle.
Change in Intrinsic Motivation for Eating Fruits and Vegetables | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  In the format of a questionnaire, participants are asked to indicate the extent to which each reason is true for them, using a 7-point scale. Why they eat fruits and vegetables (from a list of 17 reasons). Each individual question is assessed separately, so no total range is given.
Change in Intrinsic Motivation for Exercising | Baseline (Day 0), Day 30 +/- 7 days post-intervention
  In the format of a questionnaire, participants are asked to indicate the extent to which each reason is true for them, using a 7-point scale. Why they choose to exercise (from a list of 15 reasons).
Self Efficacy in Seeking Mental Health Treatment (SESMHC) | Immediately post-simulation (Day 0)
  This questionnaire consists of 9 statements. Participants are asked to rate how confident they are about each of the statements. Their responses range from 0 (no confidence) to 4 (complete confidence). The total score ranges from 0-36. The higher the score, the more confident the participant is about seeking mental health care.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Shoenthaler, EdD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Antoinette.Schoenthaler@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.